CLINICAL TRIAL: NCT02333058
Title: Clinical Phase II Trial to Describe the Safety and Efficacy of Treosulfan-based Conditioning Therapy Prior to Allogeneic Haematopoietic Stem Cell Transplantation in Paediatric Patients With Haematological Malignancies
Brief Title: Treosulfan-based Conditioning in Paediatric Patients With Haematological Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: Celerion (Industry); Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC-FludT.17/M
Record Dates: First submitted 2014-12-22; First posted 2015-01-07 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Acute Lymphoblastic Leukaemias (ALL); Acute Myeloid Leukaemias (AML); Myelodysplastic Syndromes (MDS); Juvenile Myelomonocytic Leukaemias (JMML)
Keywords: ALL; AML; MDS; JMML
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treosulfan (Experimental): Treosulfan dose per day is to be calculated by using BSA. One dose of Treosulfan per day on three consecutive days (day -6, day -5 and day -4) as intravenous (i.v.) infusion, given over 2 hours.
  Two background conditioning regimens with Treosulfan are allowed: One regimen consists of a standardised Fludarabine-containing regimen (regimen A) and the other consists of an intensified regimen with Fludarabine and ThioTEPA (regimen B). The investigator decides for each individual patient whether to treat the patient with regimen A or with regimen B.
  Treosulfan: i.v., BSA adapted: 10, 12 or 14 g/m²/day within 120 min to be administered prior to Fludarabine; Fludarabine: i.v., 30 mg/m2/day on days from -7 to -3 prior to HSCT; ThioTEPA (Regimen B): i.v., 2 x 5mg/kg/day on day -2.
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — Treosulfan dose per day is to be calculated by using BSA:
  One dose of Treosulfan per day on three consecutive days (day -6, day -5 and day -4) as intravenous (i.v.) infusion, given over 2 hours.
  Two background conditioning regimens with Treosulfan are allowed: One regimen consists of a standardised Fludarabine-containing regimen (regimen A) and the other consists of an intensified regimen with Fludarabine and ThioTEPA (regimen B). The investigator decides for each individual patient whether to treat the patient with regimen A or with regimen B.
  Treosulfan: i.v., BSA adapted: 10, 12 or 14 g/m²/day within 120 min to be administered prior to Fludarabine; Fludarabine: i.v., 30 mg/m2/day on days from -7 to -3 prior to HSCT; ThioTEPA (Regimen B): i.v., 2 x 5mg/kg/day on day -2.
  Other Names: Treograft®; Ovastat®

SUMMARY:
The primary goal of this study is to evaluate an alternative myeloablative, but reduced toxicity conditioning regimen in children, to describe the safety and efficacy of intravenous (i.v.) Treosulfan administered as part of a standardised Fludarabine-containing conditioning and to contribute to the current pharmacokinetic model to be able to finally give age (or body surface area) dependent dose recommendations. The treatment regimens given in the protocol MC-FludT.17/M are based on sufficient clinical safety and efficacy data. Considering the vital indication for allogeneic haematopoietic stem cell transplantation of the selected patient population, the risk-benefit assessment is therefore reasonably in favour of the study conduct.

DETAILED DESCRIPTION:
The protocol MC-FludT.17/M is a clinical phase II trial to describe the safety and efficacy of Treosulfan-based conditioning therapy prior to allogeneic haematopoietic stem cell transplantation (allo-HSCT) in at least 70 paediatric patients with haematological malignancies (male and female children with haematological malignant diseases as acute lymphoblastic leukaemias (ALL), acute myeloid leukaemias (AML), myelodysplastic syndromes (MDS) and juvenile myelomonocytic leukaemias (JMML), requiring myeloablative conditioning treatment with following allo-HSCT).

Treosulfan dose per day is to be calculated by using body surface area (BSA). Two background conditioning regimens with Treosulfan are allowed: One regimen consists of a standardised Fludarabine-containing regimen and the other consists of an intensified regimen with Fludarabine and ThioTEPA.

Freedom from transplant (treatment)-related mortality (TRM), defined as death from any transplant-related cause from the day of first administration of study medication until day +100 after HSCT is the primary objective of the trial.

Moreover, the current pharmacokinetic (PK) model should be contributed to be able to finally give age (or BSA) dependent dose recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Haematological malignant disease i.e. ALL, AML, MDS or JMML, indicated for allo-HSCT.
2. Indication for first allo-HSCT or second allo-HSCT due to disease relapse, graft failure, or secondary malignancy after previous HSCT.
3. Available matched sibling donor (MSD), matched family donor (MFD) or matched unrelated donor (MUD). For bone marrow (BM) and peripheral blood (PB) match is defined as 9/10 or 10/10 allele match after four digit typing in human leucocyte antigens (HLA)-A, B, C, DRB1 and DQB1.
4. Patients with ALL or AML in complete morphologic remission (blast counts <5 % in BM) and patients with MDS or JMML with blast counts < 20 % in BM at study entry.
5. Age at time of registration from 28 days to less than 18 years of age.
6. Lansky (patients aged <16 years) or Karnofsky (patients aged ≥ 16 years) performance score of at least 70 %.
7. Written informed consent of the parents/ legal guardians and patient's assent/consent according to national regulations.
8. Females of child-bearing potential or male patients' partners with child-bearing potential must use a highly effective method of contraception (pearl index < 1 %) such as complete sexual abstinence, combined oral contraceptive, hormone intrauterine contraceptive device (IUCD), vaginal hormone ring, transdermal contraceptive patch, contraceptive implant or depot contraceptive injection in combination with a second method of contraception like a condom or a cervical cap / diaphragm with spermicide or surgical sterilisation (vasectomy) in male patients or male partners during the study and at least 6 months thereafter.
9. Negative pregnancy test for females of child-bearing potential.

Exclusion Criteria:

1. Third or later allo-HSCT.
2. HSCT from haploidentical or umbilical cord blood donor.
3. Symptomatic involvement of central nervous system (CNS) at study entry.
4. Treatment with cytotoxic drugs within 10 days prior to day 7.
5. Obese paediatric patients with body mass index: weight (kg)/[height (m)]² > 30 kg/m².
6. Solid tumours (e.g. neuroblastoma, peripheral neuroectodermal tumour [PNET], Ewing sarcoma).
7. Fanconi anaemia and other deoxyribonucleic acid (DNA) breakage repair disorders.
8. Impaired liver function indicated by Bilirubin > three times the upper limit of normal (ULN) or aspartate aminotransferase/alanine aminotransferase (AST/ALT) > five times ULN, or active infectious hepatitis.
9. Impaired renal function indicated by estimated glomerular filtration rate ([GFR], according to the Schwartz formula) < 60 mL/min/1,73m2.
10. Impaired cardiac function: severe cardiac insufficiency indicated by left ventricle ejection fraction (LVEF) < 35 %.
11. Requirement for supplementary continuous oxygen.
12. Severe active infection requiring deferral of conditioning.
13. Human immunodeficiency virus (HIV) positivity.
14. Known pregnancy, breast feeding.
15. Known hypersensitivity to Treosulfan and/or Fludarabine.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2016-12-24 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Freedom from transplant (treatment)-related mortality (TRM) | from the day of first administration of study medication until day +100 after HSCT
  TRM is defined as death from any transplant-related cause

SECONDARY OUTCOMES:
Engraftment after HSCT | until engraftment
  Engraftment is defined as first of three consecutive days for each of the following four criteria:
  * a leukocyte count of more than 1 x 109/L
  * an absolute neutrophil count (ANC) of more than 0.5 x 109/L
  * a platelet count of at least 20 x 109/L in the absence of platelet transfusion
  * a platelet count of at least 50 x 109/L in the absence of platelet transfusion
Safety including early toxicity until day +100 after HSCT, serious adverse reactions (SARs) until the end of the longer-term follow-up phase | until 12 months after HSCT
  based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Hepatic sinusoidal obstruction syndrome (HSOS), lung toxicity (CTCAE term pulmonary fibrosis), hepatic toxicity and infections of any CTCAE grade (non-serious and serious) | until day +100 after HSCT
Donor-type chimerism | on day +28, day +100 and 12 months after HSCT
  The incidences of complete donor-type chimerism will be estimated as the number of patients with complete chimerism divided by the total number of patients at risk.
Non relapse mortality (NRM), transplant related mortality (TRM), graft failure rate, incidence of relapse/progression, relapse-free/progression-free survival (RFS/PFS) and overall survival (OS) | after 12 months after HSCT and until the end of the longer-term follow-up phase
  Non-relapse mortality will be defined as the probability of dying in the absence of persisting disease or previous occurrence of relapse/progression or graft failures.
  TRM is defined as the probability of dying from a transplant-related cause. The associated time span is defined as the interval from day 0 to death due to a transplant-related cause.
  The incidence of relapse/progression is defined as the probability of having relapse/progression of the underlying disease.
  Relapse-free/progression-free survival is defined as the time length between day 0 and the date of relapse/progression of the underlying disease or death due to any cause.
  OS after HSCT is defined as the probability of surviving. Survival time is defined as the time period between day 0 and the day of death due to any cause.
  Kaplan-Meier methods will be applied for estimating the probability of these parameters over time.
Incidence and severity of acute (until day +100) and chronic (until 12 months after HSCT) graft versus host disease (aGvHD/cGvHD) | until 12 months after HSCT
  The probability of grade I-IV and grade III-IV aGvHD will be estimated by cumulative incidence rates and summarised for selected time points together with their approximate 90 % confidence intervals.
  As for aGvHD, the probability of cGvHD will be estimated by cumulative incidence rates.
Use of rescue therapies including donor-lymphocyte infusions (DLIs) and further conditioning regimens | until 12 months after HSCT
PK parameters of Treosulfan and its epoxides | day -6 prior to HSCT
  The following PK parameters of Treosulfan and its epoxides will be measured: Clearance (CL); volume of distribution (Vss); terminal elimination rate constant (λz); terminal elimination half-life (t1/2); area under the concentration time curve from time zero to infinity (AUC∞); maximum observed concentration (Cmax, i.e. C end of infusion).

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Vora, MD, Prof., Principal Investigator — Great Ormond Street Hospital NHS Trust
Locations (24):
- St. Anna Children Hospital, Vienna, Austria
- University Hospital Motol, Charles University, Prague, Prague, Czechia
- Germany (13):
  - University Clinic Düsseldorf, Düsseldorf
  - University Clinic Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Essen, Essen
  - University Hospital Johann Wolfgang Goethe, Frankfurt
  - University Clinic Hamburg-Eppendorf, Hamburg
  - Medical University Hannover, Hanover
  - University Clinic Heidelberg, Heidelberg
  - University Clinic Jena, Jena
  - University Clinic München, München
  - University Clinic Münster, Münster
  - University Clinic Regensburg, Regensburg
  - University Clinic Ulm, Ulm
  - University Clinic Würzburg, Würzburg
- Italy (2):
  - Ospedale Bambino Gesu Roma, Rome
  - Ospedale Infantile Regina Margherita Torino, Turin
- Poland (4):
  - Bydgoszcz Medical University, Bydgoszcz
  - Kraków Medical University, Krakow
  - Lublin Medical University, Lublin
  - Wroclaw Medical University, Wroclaw
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Central Manchester University Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield

REFERENCES:
- [Derived] Kalwak K, Mielcarek M, Patrick K, Styczynski J, Bader P, Corbacioglu S, Burkhardt B, Sykora KW, Drabko K, Gozdzik J, Fagioli F, Greil J, Gruhn B, Beier R, Locatelli F, Muller I, Schlegel PG, Sedlacek P, Stachel KD, Hemmelmann C, Moller AK, Baumgart J, Vora A. Treosulfan-fludarabine-thiotepa-based conditioning treatment before allogeneic hematopoietic stem cell transplantation for pediatric patients with hematological malignancies. Bone Marrow Transplant. 2020 Oct;55(10):1996-2007. doi: 10.1038/s41409-020-0869-6. Epub 2020 Mar 20. PMID 32203268
- See also: sponsor's homepage — http://www.medac.de